CLINICAL TRIAL: NCT02048774
Title: Leader Partner Interactions
Acronym: LPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gregory pavela, Postdoctoral Trainee, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: X131210007
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Socioeconomic Status; Food Intake

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Social Position (Active Comparator): The investigators will randomly assign a participant to a higher social position.
  Interventions: Behavioral: Designation of Social Positioning
- Low Social Position (Experimental): The investigators will randomly assign a participant to a lower social position.
  Interventions: Behavioral: Designation of Social Positioning

INTERVENTIONS:
Behavioral: Designation of Social Positioning

SUMMARY:
Obesity is often cited as being inversely related with socioeconomic status (SES), although the mechanisms linking social status with obesity are not well understood. Dietary restraint, physical activity, and social mobility have been proposed as possible mechanisms. Although there is some evidence of SES variation in the proposed mechanisms, evidence is mixed and mostly observational. The purpose of this research is to determine if one's social position influences eating behaviors. This study will attempt to determine this using a randomized, 2 parallel arm trial to determine the effects that social hierarchy positioning has on energy intake. To prevent compromise in the integrity of data, the investigators will detail the exact treatment condition (i.e., social positioning) after the data collection period.

Based on findings from previous animal and large clinical observational studies, there are two complementary hypotheses tested in this study. First, it is hypothesized that being in a lower social position affects one's perception of food availability by making the future availability of food seem less certain. This uncertainty will lead to increased food consumption. Second, it is hypothesized that being in a position of power will lower one's food consumption, as previous research has found that individuals in power tend to east less in groups. Understanding how social position influences food intake could help improve weight loss/maintenance interventions by identifying unexpected factors that could limit the intervention's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male and female college student between the ages of 19 and 25

Exclusion Criteria:

* Those with food allergies
* Pregnant individuals

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Amount of Calories Selected and Consumed After Receiving Designation of Social Position | 1 hour after start of study

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Pavela, PhD, Principal Investigator — Postdoctoral Trainee, University of Alabama at Birmingham; Dwight Lewis, PhD, Principal Investigator — Postdoctoral Trainee, University of Alabama at Birmingham; David B Allison, PhD, Study Director — Associate Dean for Science, University of Alabama at Birmingham; Brian Wansink, PhD, Principal Investigator — Professor, Cornell University; Emily J Dhurandhar, PhD, Principal Investigator — Assistant Professor, University of Alabama at Birmingham; John Dawson, PhD, Principal Investigator — Postdoctoral Trainee, University of Alabama at Birmingham; Madeline Jeansonne, MA, Principal Investigator — Program Coordinator 1, University of Alabama at Birmingham
Locations (1):
- UAB School of Health Professions; Webb Building Rooms 503 and 504, Birmingham, Alabama, United States